CLINICAL TRIAL: NCT07009977
Title: Project BrEAtHe: Brothers, Reclaiming Emotional Awareness Tranquility Healing & Ex-istence): Disrupting Racism-related Stress, Trauma, & Problematic Substance Use
Brief Title: Project BrEAtHe: A Culturally Tailored MBSR Intervention for Young Adult Black Men
Acronym: BrEAtHe
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Phase 1 of the clinical trial completed (Delphi Panel adaptation of the MBSR trial curriculum and MBSR mhealth app development). Too few participants enrolled into the intervention (Phase 2) to continue.
Sponsor: UConn Health (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); RTI International (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Wizdom Powell, Director of Health Disparities Institute, Associate Professor of Psychiatry, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-232O-1; R34DA054412 (NIH)
Record Dates: First submitted 2024-02-16; First posted 2025-06-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Abuse; Substance Abuse; Post Traumatic Stress Disorder
Keywords: Black Men; Mindfulness-Based Stress Reduction; Substance Use; Alcohol Use; Prevention; Ecological Momentary Assessment
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Stress Disorders, Post-Traumatic; Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group based MBSR training with BrEAtHe App (No Feedback) (Experimental): self-guided mHealth app only
  Interventions: Behavioral: self-guided mHealth app only
- Group based MBSR training with BrEAtHe App (Feedback) (Experimental): self-guided mHealth app + 'real-time' feedback.
  Interventions: Behavioral: self-guided mHealth app + 'real-time' feedback

INTERVENTIONS:
Behavioral: self-guided mHealth app only — Mindfulness based stress reduction
  Arms: Group based MBSR training with BrEAtHe App (No Feedback)
Behavioral: self-guided mHealth app + 'real-time' feedback — Mindfulness based stress reduction with mobile app feedback
  Arms: Group based MBSR training with BrEAtHe App (Feedback)

SUMMARY:
The purpose of this study is to create a program focused on mindfulness and stress reduction specifically tailored to young adult Black males.

DETAILED DESCRIPTION:
Project Brothers reclaiming Emotional Awareness, tranquility, Healing, and Ex-istence (BrEAtHe) is a research study to create a program focused on mindfulness and stress reduction specifically tailored to young adult Black males (18 to 29 years old) residing in Durham, NC and in Hartford, CT. The investigators plan to use a mobile app on a cell phone to better understand 'real-time' feedback of experiences of stress due to racism. The investigators are interested in learning about the recruitment and retention of Black males participating in mindfulness based practices. The investigators are also interested in receiving feedback about options to modify and scale a Mindfulness Based Stress Reduction intervention and its preliminary effects on reducing physical and emotional stress reactions and poor coping mechanisms like marijuana and alcohol use linked to everyday racism and discrimination.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-29
* Ethnicity: non-Hispanic Black
* Gender: Male
* does not meet the DSM-V criteria for substance use disorder or dependence or severe post-traumatic stress disorder (PTSD);
* Neighborhood Inclusion Criteria: must live in a high VAOD neighborhood in Durham County, NC, or North Hartford Promise Zone, CT and have resided in the selected neighborhood for at least 6 months.

Exclusion Criteria:

* non-English speakers,
* meet the DSM-V criteria for substance use disorder or dependence or severe post-traumatic stress disorder (PTSD);
* women;
* men of other racial/ethnic groups;
* neighborhood outside of high VAOD neighborhood in Durham County, NC or North Hartford Promise Zone, CT.

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Daily Marijuana use levels | immediately before and after the intervention
  Daily marijuana use will be assessed with ecological momentary assessment (EMA). Participants will be asked to respond to random digital prompts on a handheld mobile device about recent substance use. Questions will include "Within the past hour, have you: (used marijuana)?" The response anchors for these questions will be "NO" or "YES." To classify alcohol or marijuana use confirmed with a "YES" response as problematic, The Drug Abuse Screening Test (DAST-10) will be administered. A separate summed score will be created for alcohol and marijuana use levels based on DSM-V criteria with higher scores indicating more problematic alcohol or marijuana use.
Daily Alcohol use levels | immediately before and after the intervention
  Daily alcohol use will be assessed with ecological momentary assessment (EMA). Participants will be asked to respond to random digital prompts on a handheld mobile device about recent alcohol use (drank alcohol)?" The response anchors for these questions will be "NO" or "YES." To classify alcohol or marijuana use confirmed with a "YES" response as problematic, The Alcohol Use Disorders Identification Test (AUDIT-C) will be administered. A separate summed score will be created for alcohol and marijuana use levels based on DSM-V criteria with higher scores indicating more problematic alcohol or marijuana use.
Daily Racism-Related and General Stress | immediately before and after the intervention
  Daily racism-related and general stress will be assessed with questions about asked the occurrence and impact of stress related to general experiences (i.e., had money troubles; argued with spouse or partner; had transportation problems) and those attributed to experiences of everyday racism (i.e., been followed by police officers or neighborhood security patrols because of your race). The response anchors for these questions will be "NO" or "YES." The impact of these experiences will be rated on a 5-point scale (1=not at all to 5=very stressful). Higher scores on these measures indicate more frequent and impactful stress experiences. Participants will also be asked to initiate an entry when they experience an impactful everyday racism or general stress experience at times not coinciding with Random Digital Prompts or RDPs (also called event-contingent entries)

SECONDARY OUTCOMES:
Trauma Symptomatology | immediately before and after the intervention
  Trauma symptomatology will be assessed with items from a shortened, 7-item version of the Civilian Version of the Post-Traumatic Stress Disorder Checklist for the Diagnostic Statistical Manual 5 or (PCL-5). This scale uses a dichotomous scoring scheme of 1 "yes" or 0 "no" for each item. Higher scores will indicate the presence of higher trauma symptomatology.
Affect Regulation (i.e., emotion suppression) | immediately before and after the intervention
  Investigators will assess affect regulation using the 10-item Emotion Regulation Questionnaire (ERQ) continuous measure assesses individual differences in the habitual use of emotion suppression and cognitive reappraisal. Consistent with previous EMA research, participants will be asked to indicate their affect regulation strategies (emotion suppression vs. reappraisal) for experiences they rate as highly stressful (3 or more rating) by responding to questions derived from the ERQ described above, "Try to remember how you responded to your feelings about this experience; Did you keep your feelings about the experience to yourself, or try to think about your feelings and the experience in a different way?" Higher scores indicate a higher participant use of and reliance on emotion suppression.
Stress Reactivity (i.e., Heart Rate Variability (HRV)) | immediately before and after the intervention
  Heart Rate Variability (HRV) will be assessed with a Faros monitor, which captures ECG at a 1000 Hz sampling frequency. A mechanism will be set on this device to assure synchrony between physiological and behavioral data. HRV monitoring will be conducted on Day 1 and post intervention for 15 minutes each.
Acceptability (User Satisfaction, Intent to Continue, Perceived Appropriateness, Fit, & Demand of Use) | immediately after the intervention
  Acceptability will be assessed with quantitative survey measures (user satisfaction, intent to continue, perceived appropriateness, fit within disadvantaged neighborhood settings and among young adult Black males, and demand or use of BrEAtHe intervention strategies and app).

OTHER OUTCOMES:
Feasibility (Recruitment, Daily Completion, & Drop-out Rates) | immediately after the intervention
  Feasibility will be assessed by examining logged days of training derived from attendance records and app usage (the number of participant-initiated and app-initiated practices).
Perceptions of Delivery modalities | immediately after the intervention
  Post-intervention questionnaires will be used to gather insights about young adult Black men's intervention participation experiences and perceptions of the delivery modalities.
Changes in Daily Substance Use | Immediately after the 8-9 week intervention
  Investigators will explore whether participation in the mindfulness based intervention led to reductions in daily non-problematic and problematic usage of alcohol or marijuana as determined by criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). A separate summed score will be created from dichotomous responses ("YES" or "NO") to questions about the frequency and impact of daily alcohol and marijuana use with higher scores indicating more frequent and problematic alcohol or marijuana use.
Changes in Daily Stress-Affective and Trauma Response | Immediately after the 8-9 week intervention
  Investigators will explore whether the intervention led to reductions in intermediary stress, trauma symptomatology, emotion regulation, and Heart Rate Variability (HRV). Investigators will examine changes between baseline and post-intervention scores on the PCL-5 (trauma symptomatology), ERQ (emotion regulation), and HRV assessments (Faros monitoring).

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided